CLINICAL TRIAL: NCT03081754
Title: Study of Placental Bed of Growth Restricted Fetuses: Correlation of Doppler Velocimetries of Uterine and Umbilical Arteries With Placental Pathology
Brief Title: Correlation of Uterine and Umbilical Arteries Doppler With Placental Pathology in IUGR
Status: Completed | Type: Observational
Sponsor: Ahmed Maged (Other)
Responsible Party: Sponsor-Investigator, Ahmed Maged, Assistant professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 160
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The general shapes of placentas were assessed and weightedby trimming the membranes and umbilical cord. The diameters and thickness of placentas were noted cord insertion site. The maternal surface at a distance of 1-2 cm in bread loaf manner and examined for the pale areas. Whole thickness villous tissue blocks were obtained from three zones ;central, peripheral and intermediate zones
  Placental bed biopsies were obtained at Caesarean sections .. The specimens were fixed in buffered formalin. The tissues were processed and stained with Haematoxlyin and Eosin. Microscopic study of placenta was carried out utilizing a set of standard criteria for villous and intervillous lesions . For studying these criteria 8 random microscopic fields were chosen and 100 villi were counted in each field
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IUGR: Fifty women with intrauterine growth restricted fetuses were included in the study. Gestational age was based on the precisely dated last menstrual period and ultra-sonographic examination of crown-rump length in the first trimester. Intrauterine growth restriction was diagnosed when fetal abdominal circumference was more than two standard deviations below the mean for gestational age and also confirmed by the serial assessment of the fetal growth parameters (Chitty and Altman, 1999). Detailed obstetric history was available for each patient. Caesarean sections were performed on clinical grounds
  Interventions: Radiation: Doppler velocimetry
- control group: Twenty five uneventful pregnancies with appropriate for gestational age fetuses are selected as control. Obstetric history Doppler results and placenta were examined for any remarkable pathology. Caesarean sections were performed on clinical grounds. The indications for Caesarean section of the controls, which were tried to be at equivalent gestational ages with the study group, were presentation abnormalities or previous Caesarean section
  Interventions: Radiation: Doppler velocimetry

INTERVENTIONS:
Radiation: Doppler velocimetry — Doppler studies were performed within the last week before delivery using a 3.5-Mhz transducer, all measurements were performed with the mothers in a semi recumbent position. Color-flow imaging was used to visualize the ascending branch of the uterine arteries. Pulsed Doppler velocimetry was performed with a sample volume of 5 mm.

SUMMARY:
When indicated, a conservative management plan of IUGR was undertaken. Doppler studies were performed within the last week before delivery The results of Umbilical artery (UA) Doppler velocimetry were categorized as normal , increased , absent, and reversed . Patients were admitted for close surveillance in the case of worsening of maternal or fetal conditions (e.g. absent or reversed UA blood flow, and severe preeclampsia).

Tissue samples The general shapes of placentas were assessed. The collected placentas were weighed by trimming the membranes and umbilical cord. Then the diameters and thickness of placentas were noted. The position of insertion of umbilical cord on the fetal surface of placenta was observed. Transverse cuts were made through the maternal surface at a distance of 1-2 cm in bread loaf manner and examined for the pale areas. All placentas were immersed in 10% formalin overnight and examined on the next day. For each placenta, blocks containing cord, membrane and full thickness of villous tissue were prepared. Whole thickness villous tissue blocks were obtained from three zones, i)central zone ii) peripheral zone and iii) intermediate zone between the first two zones, so as to include all areas of placenta.

Placental bed biopsies were obtained at Caesarean sections with direct visualization of the placental site. Biopsies of at least 1cm were taken. The specimens were fixed in buffered formalin. The tissues were processed and stained with Haematoxlyin and Eosin. Microscopic study of placenta was carried out utilizing a set of standard criteria for villous and intervillous lesions

Immunohistochemistry Expression of VEGF and CD34 was analyzed in 75 (50 placenta of IUGR and 25 of control) placental villous tissues.

Immunostaining was performed by the streptavidin-biotin-peroxidase method. Evaluation of immunohistochemical staining To determine the MVD, the stained placental vasculature. Tissue sections were initially screened microscopically at low power (100×) to identify the areas of highest vascularization ("hot spots").

Evaluation of immunohistochemical staining of VEGF:

DETAILED DESCRIPTION:
When indicated, a conservative management plan of IUGR was undertaken according to a defined protocol including antenatal visits, ultrasound surveillance. The frequency of fetal surveillance was assessed at each visit according to the maternal and fetal conditions.

Doppler studies were performed within the last week before delivery using a 3.5-Mhz transducer, color-flow mapping, and a 50-Hz high-pass filter; all measurements were performed with the mothers in a semi recumbent position. Color-flow imaging was used to visualize the ascending branch of the uterine arteries. Pulsed Doppler velocimetry was performed with a sample volume of 5 mm.

A minimum of three separate recordings was taken for each examination. The wave contour of the uterine arteries was studied for the presence of a diastolic notch from which the systolic/end-diastolic (S/ D) ratio was calculated. Abnormal uterine velocimetry was defined as an average of (left and right) S/ D ratio and by the bilateral presence of diastolic notching. Umbilical artery waveform was measured from free-floating loop of cord during fetal quiescence. The pulsatility index (PI) (maximum velocity - minimum velocity/ mean velocity) was calculated and the average of three measurements was used. An abnormal umbilical artery PI was defined as standard deviations above the mean for gestational age based reference standards (Chitty and Altman, 1999).

The results of Umbilical artery (UA) Doppler velocimetry were categorized as normal (end-diastolic velocity <90th percentile of our reference curve), increased (end-diastolic velocity ≥90th percentile), absent, and reversed (Madazil R et al., 2002) Patients were admitted for close surveillance in the case of worsening of maternal or fetal conditions (e.g. absent or reversed UA blood flow, and severe preeclampsia). Preeclampsia was defined according to standard criteria (Arduini D et al, 2002).

Tissue samples The general shapes of placentas were assessed. The collected placentas were weighed by trimming the membranes and umbilical cord. Then the diameters and thickness of placentas were noted. The position of insertion of umbilical cord on the fetal surface of placenta was observed. Transverse cuts were made through the maternal surface at a distance of 1-2 cm in bread loaf manner and examined for the pale areas. All placentas were immersed in 10% formalin overnight and examined on the next day. For each placenta, blocks containing cord, membrane and full thickness of villous tissue were prepared. Whole thickness villous tissue blocks were obtained from three zones, i)central zone ii) peripheral zone and iii) intermediate zone between the first two zones, so as to include all areas of placenta.

Placental bed biopsies were obtained at Caesarean sections with direct visualization of the placental site. Biopsies of at least 1cm were taken. The specimens were fixed in buffered formalin. The tissues were processed and stained with Haematoxlyin and Eosin. Microscopic study of placenta was carried out utilizing a set of standard criteria for villous and intervillous lesions (Kotigwar S et al 2011). For studying these criteria 8 random microscopic fields were chosen and 100 villi were counted in each field and studied for the presence of following criteria:

1. Syncytial knots >30% in one field
2. Fibrinoid necrosis >5% in one field
3. Placental infarction >5% in one field Intervillous space

a) Chorangiosis b) Perivillous fibrinoid deposition >5% in one field c) Infarctions d) Presence of calcification. e) Thickened hylinosed blood vessels For statistical purpose such changes are labeled as "Abnormal placenta"

Immunohistochemistry Expression of VEGF and CD34 was analyzed in 75 (50 placenta of IUGR and 25 of control) placental villous tissues. Samples (1.5 × 1.5 × 1 cm in diameter) taken from the maternal surface of each placenta; infarct areas were excluded from the study. All tissues were fixed in formalin, embedded in paraffin, and cut into 5-μm-thick sections, which were collected on slides coated with poly-L-lysine. After the paraffin was removed, the sections were rehydrated.

Immunostaining was performed by the streptavidin-biotin-peroxidase method. Endogenous peroxidase activity was blocked using 3% hydrogen peroxide. Antigen retrieval was carried out in a microwave oven for 15 minutes in 10 nM citrate buffer (pH 6.0) for VEGF. The sections were incubated at room temperature for one hour with EP1176Y rabbit polyclonal antibodies reactive with VEGF (1:100; Genova, Spain), CD34 mouse monoclonal antibodies Ventana. USA). After washing in phosphate-buffered saline with Tween-20, the tissues were incubated with a biotin-conjugated secondary antibody and then with a biotin-streptavidin complex for 30 min at room temperature. Reactions were visualized with 3,3-diaminobenzidine tetrahydrochloride (DAB). Sections were counterstained with hematoxylin, rinsed, and mounted.

Evaluation of immunohistochemical staining

Evaluation of immunohistochemical staining of CD34:

Microvessel Density Determination

The most popular method to study the angiogenic activity in a tissue is to count the number of microvessels per unit area of tissue section, known as the microvessel density (MVD). (Hasan J et al, 2002) To determine the MVD, the stained placental vasculature. Tissue sections were initially screened microscopically at low power (100×) to identify the areas of highest vascularization ("hot spots"). Five high-power (400×) fields were then chosen randomly, and the number of microvessels in each high-power field (0.09 mm2) was counted for each sample with the use of an ocular grid. MVD for each sample was taken as the mean of the five values obtained. (Mustafa G et al, 2012)

Evaluation of immunohistochemical staining of VEGF:

The intensity and localization of the staining reaction in chorionic villous stromal cells, vascular smooth muscle cells, villous vascular endothelial cells, cytotrophoblasts, syncytiotrophoblasts, and extravillous trophoblasts was evaluated. Immunoreactivity for antibodies was scored using a semi-quantitative scale for intensity of staining: 0 negative, no staining; 1+ weak positive; 2+ moderately positive; 3+ strongly positive. (Barut F et al, 2010)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational age 28-34 weeks fetal growth below 5th percentile

Exclusion Criteria:

* Pregnancies with known vascular maternal disease (chronic hypertension, autoimmune diseases, and diabetes) fetuses with structural abnormalities twins

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 1. Group 1 ( control group) :
     Twenty five uneventful pregnancies with appropriate for gestational age fetuses are selected as control.
  2. Group 2:
  Fifty women with intrauterine growth restricted fetuses were included in the study. Gestational age was based on the precisely dated last menstrual period and ultra-sonographic examination of crown-rump length in the first trimester. Caesarean sections were performed on clinical grounds
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Doppler correlation with placental pathology | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes